CLINICAL TRIAL: NCT02215239
Title: Development of Workplace Physical Activity Promotion Models in Taiwan
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 201310041RINA
Record Dates: First submitted 2014-08-11; First posted 2014-08-13 (Estimated); Last update posted 2015-03-17 (Estimated); Status verified 2015-03

CONDITIONS: Occupational Health
Keywords: health lifestyle; health promotion; occupational health; Work site health promotion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Working type A & Workplace intervention (Experimental): Participants: Workers tend to be seated during work hours. Intervention: WHO Healthy Workplace Framework and Model. Duration: 16 weeks.
  Interventions: Behavioral: Workplace intervention
- Working type A & Usual care (No Intervention): Participants: Workers tend to be standing during work hours. Intervention: Usual care. Duration: 16 weeks.
- Working type B & Workplace intervention (Experimental): Participants: Workers tend to be standing during work hours. Intervention: WHO Healthy Workplace Framework and Model. Duration: 16 weeks.
  Interventions: Behavioral: Workplace intervention
- Working type B & Usual care (No Intervention): Participants: Workers tend to be standing during work hours. Intervention: Usual care. Duration: 16 weeks.

INTERVENTIONS:
Behavioral: Workplace intervention — WHO Healthy Workplace Framework and Model. The intervention plan is to implement a cyclic or iterative process recommended by WHO. The process includes eight steps: (1) Mobilize; (2) Assemble; (3) Assess; (4) Prioritize; (5) Plan; (6) Do; (7) Evaluate; (8) Improve. We focus on different phases of exercise and prescribe individualized physical activity program.
  Arms: Working type A & Workplace intervention; Working type B & Workplace intervention

SUMMARY:
The purpose of this study is to investigate the effectiveness of intervention applying WHO Healthy Workplace Framework and Model to enhance the level of physical activity on employees. This research is an experimental intervention study recruiting two working types in four workplaces. Two working types are: (1) Working type A: Workers tend to be seated during work hours. Two telecommunications enterprises will respectively stand for the experiment group and the control group. (2) Working type B: Workers tend to be standing during work hours. Likewise, two different enterprises will respectively stand for the experiment group and the control group. Purposive sampling method will be used to select the experiment group. The intervention plan is to implement a cyclic or iterative process recommended by WHO.

DETAILED DESCRIPTION:
Several evidences have shown that regular physical activity could benefit not only to a healthy lifestyle, but also reduce mortality rate. However, the number of people who perform regular physical activity are still in a low proportion of world population. In Taiwan, people are mostly inactive and have low level of physical activity at their workplaces. Therefore, developing a healthy workplace could encourage employees to get into the habit of regular exercise, relieve stress, improve interaction of social activity and build a healthy life style. Meanwhile, regular exercise could improve coherence, morale and higher satisfaction, productive efficiency, corporate image and competitiveness. Previous studies have shown inconsistent effects in promoting physical activity in the workplace. Therefore, determining the effects of comprehensive model using in interventions at workplaces is needed. . The purpose of this study is to investigate the effectiveness of intervention applying WHO Healthy Workplace Framework and Model to enhance the level of physical activity on employees. This research is an experimental intervention study recruiting two working types in four workplaces. Two working types are: (1) Working type A: Workers tend to be seated during work hours. Two telecommunications enterprises will respectively stand for the experiment group and the control group. (2) Working type B: Workers tend to be standing during work hours. Likewise, two different enterprises will respectively stand for the experiment group and the control group. The intervention plan is to implement a cyclic or iterative process recommended by WHO. The process includes eight steps: (1) Mobilize; (2) Assemble; (3) Assess; (4) Prioritize; (5) Plan; (6) Do; (7) Evaluate; (8) Improve. By gaining the commitment from the highest authority in the enterprise and communicated to all workers and their representatives, we will be able to assemble a Healthy Workplace Team who will work on implementing change in the workplace. As well as assembling the Team, it is also essential to assemble other resources that will be required, such as locations, time, budgets or working supplies, to ensure the committee has the resources necessary to do the work. Assessments on both the present situation of the enterprise and the present situation with respect to the health of workers are required in order to set priorities among the many issues identified. When developing a health plan, we focus on different phases of exercise and prescribe individualized physical activity program., in the mean while, the power of social learning and environmental support are critical in making a sustainable improvement in the workplace. The details of the actions to be taken may contain educational workshop, pedometer using, setting fixed period of time for physical activities, providing excellent health and fitness improvement prize, email and text reminder about exercise information, holding outdoor physical activities on a regular time schedule for employee, and propagating internal and external resources. Re-evaluation and modification will be performed at the end of 16-weeks intervention, and then the second year's study will be planned and designed. In the present study, before intervention, we will require a confidential survey and health risk assessments about personal health condition base on employees will. The assessments include basic data and medical record, level of physical activity, health-related fitness, sleep quality and daytime sleepiness, depression scale, exercise stages, self-evaluation of fitness and exercise capacity, self-efficacy in exercise, SmartIn(SI) system, and working performance evaluation. The purpose of the study is to access the effect of implementing The WHO Healthy Workplace Framework and Model on different working types in different workplaces, by developing method that address the physical and psychosocial working environments, as well as promoting workers' health and creating health-promoting working environments, the result is expected to provide better information for the Health Promotion Administration in future policy-making.

ELIGIBILITY:
Inclusion criteria:

* Workers tend to be seated or standing during work hours.
* Basic capability to read or verbal communication in Chinese.

Exclusion criteria:

* No other critical diseases or unstable cardiopulmonary disease, diabetes, hypertension or neurological diseases.
* No pregnancy.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2014-01; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Change of health-related physical fitness from baseline to 16-week | 16 weeks
  Health-related physical fitness including:
  1. body composition (body weight, height, waist and hip circumferences)
  2. flexibility (sit-to-reach, cm)
  3. muscle strength (grip strength of dominant hand, kg)
  4. muscle endurance (sit-up in one minute, times/min)
  5. cardiopulmonary endurance (stepping in three minutes, heart rate and physical exercise index)

SECONDARY OUTCOMES:
Change of physical activity from baseline to 16-week | 16 weeks
  Using 7-Day Physical Activity Recall questionnaire and actigraph to investigate level of physical activity in the participants
Change of sleep quality from baseline to 16-week | 16 weeks
  Using Pittsburgh Sleep Quality Index, Epworth Sleepiness Scale, and actigraph to investigate sleep quality in the participants
Change of depression symptoms from baseline to 16-week | 16 weeks
  Using Center for Epidemiologic Studies Depression Scale to investigate level of depression in the participants
Change of stress from baseline to 16-week | 16 weeks
  Using SmartIn system to investigate level of psychological stress in the participants

CONTACTS AND LOCATIONS:
Overall Officials: Meng-Yueh Chien, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan